CLINICAL TRIAL: NCT01879098
Title: Evaluation of the Effect of 3 Probiotic Strains on Bile Acids, Satiety, and Inflammation in Healthy, Middle-aged Adults: a Randomized, Double-blinded, Placebo-controlled Study
Brief Title: The Effect of 3 Probiotic Strains on Bile Acids, Satiety, and Inflammation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB# 70-2013
Record Dates: First submitted 2013-06-12; First posted 2013-06-17 (Estimated); Last update posted 2014-07-10 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
Keywords: probiotics; inflammation; bile; hunger; satiety
MeSH Terms: conditions — Inflammation | interventions — bificin C6165, Bifidobacterium animalis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo will be taken once daily for 6 weeks by every subject at some point in the study (crossover design).
  Interventions: Dietary Supplement: Placebo
- Probiotic: Bacillus subtilis (Experimental): Bacillus subtilis will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Probiotic: Bacillus subtilis
- Probiotic: Lactobacillus plantarum (Experimental): Lactobacillus plantarum will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Lactobacillus plantarum
- Probiotic: Bifidobacterium animalis (Experimental): Bifidobacterium animalis will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Interventions: Dietary Supplement: Bifidobacterium animalis

INTERVENTIONS:
Dietary Supplement: Probiotic: Bacillus subtilis — Bacillus subtilis will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Other Names: Bacillus subtilis R0179
  Arms: Probiotic: Bacillus subtilis
Dietary Supplement: Lactobacillus plantarum — Lactobacillus plantarum will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Other Names: Lactobacillus plantarum HA-119
  Arms: Probiotic: Lactobacillus plantarum
Dietary Supplement: Bifidobacterium animalis — Bifidobacterium animalis will be taken as a capsule once daily for 6 weeks by subjects in the group receiving this supplement (group is unknown, double-blinded).
  Other Names: Bifidobacterium animalis subsp. lactis LAFTI B94
  Arms: Probiotic: Bifidobacterium animalis
Dietary Supplement: Placebo — Placebo will be taken once daily for 6 weeks by every subject at some point in the study (crossover design).
  Arms: Placebo

SUMMARY:
The purpose of this research study is to determine whether a probiotic can change the way bile is used by the body. The investigators will also look at the effect of the probiotic on your intestinal health.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled crossover study. After obtaining informed consent, healthy, middle-aged adults with a larger waist circumference (n=30/probiotic cross with n=90 total/study) will be randomized to one of four groups: Bacillus subtilis, Lactobacillus plantarum, Bifidobacterium animalis subsp. lactis, or placebo. Participants will consume 1 capsule per day of probiotic or placebo for 6 weeks. After a 4-week washout period, participants will be crossed to the other treatment (i.e., probiotic to placebo or placebo to probiotic).

Participants will complete daily questionnaires throughout the intervention period, and one week before and after each intervention period. Blood samples will be collected at the baseline and final time points (±3 days) of each intervention. Stool samples will be collected during the pre-baseline and final weeks of each intervention. Dietary intake will be assessed weekly during each intervention period. Gastrointestinal symptoms and physical activity questionnaires will be completed weekly during each intervention period and also the weeks before and after each intervention period.

ELIGIBILITY:
Inclusion Criteria

To participate in the study you must:

* Be 35-65 years of age.
* Have a waist circumference > 102 cm (40 in) for males, and > 88 cm (35 in) for females.
* Be willing and able to complete the Informed Consent Form in English.
* Be available for 18 consecutive weeks to participate in this study.
* Be willing and able to complete daily and weekly questionnaires regarding general wellness, bowel function, gastrointestinal symptoms, physical activity level, and dietary intake.
* Be willing to provide 4 blood samples and 4 stool samples.
* Be willing to maintain your regular level of physical activity and your diet for 18-week study.
* Be able to take the study supplement without the aid of another person.
* Be willing to discontinue consumption of fermented foods or probiotics (e.g., yogurts with live, active cultures or supplements).
* Be willing to provide a social security number (SS#) to receive study payment. Note: the subject can still participate if unwilling to provide SS#, but no financial reimbursement can be provided.

Exclusion Criteria:

To participate in the study you must NOT:

* Fail to meet any of the criteria I mentioned above.
* Consume >20 g fiber daily, according to the Block Fiber Screener.
* Be taking any statins or cholesterol-lowering prescription drugs now, or within the last 6 months.
* Be currently taking any constipation or diarrhea on a regular basis.
* Be currently taking any systemic corticosteroids, androgens (such as testosterone), or large doses of anti-inflammatory drugs (i.e., aspirin in doses >600 mg/d) on a regular basis.
* Have used plant sterols, n-3 fatty acids, fish oil, soy protein, soluble oat fiber, psyllium seed husk or other cholesterol-lowering supplements within the last 3 months.
* Have received antibiotic therapy or a colonoscopy in the past two months.
* Currently be treated for or have any of the following physician-diagnosed diseases or conditions: HIV/AIDS; immune modulating diseases (autoimmune disease, hepatitis, cancer); kidney disease; pancreatitis; pulmonary disease; hepatic or biliary disease; or gastrointestinal diseases/conditions such as diverticulitis, ulcerative colitis, Crohn's disease, Celiac disease, short bowel disease, ileostomy, colostomy, but not including Gastroesophageal Reflux Disease (GERD); or have a central venous catheter.
* Taking medications for type 1 or type 2 diabetes.
* Be physically active or very physically active. Active = typical daily living activities PLUS at least 60 minutes of daily moderate activity. Very active = typical daily living activities PLUS at least 60 minutes of daily moderate activity, PLUS an additional 60 minutes of vigorous activity OR 120 minutes of moderate activity.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2013-08; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Difference in deconjugated bile acids in the blood | Baseline #1 (Week 1) to Week 8 and Baseline #2 (Week 11) to Week 18
  Levels of deconjugated bile acids in the stool and in the blood will be compared between treatment periods for each subject/group.

SECONDARY OUTCOMES:
Satiety and glucose metabolism | Baseline #1 (Week 1) to Week 8 and Baseline #2 (Week 11) to Week 18
  Levels of hormones associated with hunger, satiety and glucose metabolism in the blood will be compared between treatment periods for each subject/group. Daily questionnaires will also assess hunger/satiety.

OTHER OUTCOMES:
Inflammatory status | Baseline #1 (Week 1) to Week 8 and Baseline #2 (Week 11) to Week 18
  Levels of inflammatory markers in the blood will be compared between treatment periods for each subject/group.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Derived] Culpepper T, Rowe CC, Rusch CT, Burns AM, Federico AP, Girard SA, Tompkins TA, Nieves C Jr, Dennis-Wall JC, Christman MC, Langkamp-Henken B. Three probiotic strains exert different effects on plasma bile acid profiles in healthy obese adults: randomised, double-blind placebo-controlled crossover study. Benef Microbes. 2019 May 28;10(5):497-509. doi: 10.3920/BM2018.0151. Epub 2019 May 15. PMID 31090458